CLINICAL TRIAL: NCT04777032
Title: The Danish Comorbidity in Liver Transplant Recipients Study (DACOLT) - a Non-interventional Prospective Observational Cohort Study
Brief Title: The Danish Comorbidity in Liver Transplant Recipients Study
Acronym: DACOLT
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Susanne Dam Nielsen, MD, DMSc, Professor, MD, DMSc, Rigshospitalet, Denmark
Other Study IDs: Sponsor1 - Rigshospitalet
Record Dates: First submitted 2021-02-16; First posted 2021-03-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplantation; Comorbidities and Coexisting Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biochemical analyses including fasting insulin and fasting blood glucose. Blood will be collected for a research biobank, and peripheral blood mononuclear cells, serum and plasma will be stored for further analyses of inflammation markers (chemokines, cytokines, soluble surface markers), coagulation markers (standard and functional platelet aggregation test), simulation assays and flowcytometry of PBMC, endothelial function markers (asymmetric dimethylarginine (ADMA), syndecan-1, trombomodulin and sE-selectin), markers of microbial translocation and bacterial degradation (sCD14, lipopolysaccharide, trimethylamine N-oxide), markers of lung tissue (alpha-1-antitrypsine, endothelin-1), liver markers (hyaluronic acid and fibrosis markers) and metabolomics and multiomics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Liver transplant recipients: All liver transplant recipient in Denmark aged 20-100 years will be eligible for inclusion in the DACOLT study. Inclusion requires the individual to be able to understand the study information in either Danish or English and to be able to provide an informed consent.
- Control group 1_CGPS: The Copenhagen General Population Study (CGPS) is an ongoing observational population study with more than 110.000 participants from the greater Copenhagen area. All residents in the greater Copenhagen area > 40 years and 25% of 20-40 years old are invited to participate in the study and in follow-up examinations every decade. A random sample of 10.000 participants aged ≥ 40 years had a contrast enhanced CT of the chest including CT angiography of the heart performed. Of these, 6500 had a contrast enhanced CT of the abdomen.
- Control group 1_CCHS: The Copenhagen City Heart Study (CCHS) includes a random population sample included from the greater Copenhagen area. Health surveys have been repeated 5 times between 1976 and 2015. Almost 4000 participants were randomly selected for echocardiography.

SUMMARY:
Background:

Liver transplantation is the only curative treatment for patients with end-stage liver disease. Short-term survival has improved due to improved surgical techniques and greater efficacy of immunosuppressive drugs. At present, the 10-year survival after liver transplantation is 60%, but long-term survival has not improved to the same extent the short-term survival. In addition to liver- and transplant-related causes, comorbidities such as cardiovascular, pulmonary, renal, and metabolic diseases have emerged as leading causes of morbidity and mortality in liver transplant recipients.

The objective of this study is to assess the burden of comorbidities and identify both liver- and transplant-related risk factors as well as traditional risk factors that contribute to the pathogenesis of comorbidity in liver transplant recipients.

Methods/design:

The DACOLT study is an observational, longitudinal study. The investigators aim to include all adult liver transplant recipients in Denmark. Participants will be matched by sex and age to controls from the Copenhagen General Population Study (CGPS) and the Copenhagen City Heart Study (CCHS). Physical and biological measures including blood pressure, ancle-brachial index, spirometry, exhaled nitric oxide, electrocardiogram, transthoracic echocardiography, computed tomography (CT) angiography of the heart, unenhanced CT of chest and abdomen and blood samples will be collected using uniform protocols in participants in CGPS, CCHS and DACOLT. Blood samples will be collected and stored in a research biobank. Follow-up examinations at regular intervals up to 10 years of follow-up are planned.

Discussion:

There is no international consensus standard for optimal clinical care or monitoring of liver transplant recipients. The study will determine prevalence, incidence and risk factors for comorbidity in liver transplant recipients and may be used to provide evidence for guidelines on screening and long-term treatment and thereby contribute to improvement of the long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplanted
* age between 20 and 100 years
* be able to understand the study information in either Danish or English and to be able to provide an informed consent

Exclusion Criteria:

* none

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All liver transplanted individuals in Danmark.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2033-01-01 (Estimated); Study Completion 2043-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of coronary artery disease | Baseline cross-sectional data
  Assessed by coronary CT angiography
Change in Coronary artery disease | 10 years follow-up
  Assessed by coronary CT angiography
Cardiac function | Baseline cross-sectional data
  Determined by transthoracic echocardiography
Change in Cardiac function | 10 years follow-up
  Determined by transthoracic echocardiography
Cardiac structure | Baseline cross-sectional data
  Determined by transthoracic echocardiography
Change in cardiac structure | 10 years follow-up
  Determined by transthoracic echocardiography
Cardiac structure | Baseline cross-sectional data
  Assessed by cardiac computed tomography (CT)
Change in Cardiac structure | 10 years follow-up
  Assessed by cardiac computed tomography (CT)
Cardiac function | Baseline cross-sectional data
  Assessed by cardiac computed tomography (CT)
Change in Cardiac function | 10 years follow-up
  Assessed by cardiac computed tomography (CT)
Dynamic lung function indices assessed by spirometry | Baseline cross-sectional data
  FVC and FEV1 assessed by spirometry
Change in Dynamic lung function indices assessed by spirometry | 10 years follow-up
  FVC and FEV1 assessed by spirometry
Renal function | Baseline cross-sectional data
  Estimated glomerular filtration rate
Change in Renal function | 10 years follow-up
  Estimated glomerular filtration rate
Metabolic diseases | Baseline cross-sectional data
  Prevalence of Diabetes
Metabolic diseases | 10 years follow-up
  Change in Diabetes
Metabolic diseases | Baseline cross-sectional data
  Prevalence of Dyslipidaemia
Metabolic diseases | 10 years follow-up
  Change in Dyslipidaemia

SECONDARY OUTCOMES:
Prevalence of Depression | Baseline cross sectional data
  Major Depression Inventory (MDI): A depression questionnaire. The questionnaire consists of the ten symptoms contained in the World Health Organization WHO's depression demarcation. The patient's completed questionnaire is scored using a scoring key.
  When MDI is used as a rating scale in the same way as the Hamilton scales, then the sum of the ten questions indicates the degree of depression. The theoretical score range is from 0 (no depression) to 50 (maximum depression).
  Mild depression: MDI total score from 21 to 25 Moderate depression: MDI total score from 26 to 30 Severe depression: MDI total score of 31 or higher
Change in Depression | 10 years follow-up
  Major Depression Inventory (MDI): A depression questionnaire. The questionnaire consists of the ten symptoms contained in the World Health Organization WHO's depression demarcation. The patient's completed questionnaire is scored using a scoring key.
  When MDI is used as a rating scale in the same way as the Hamilton scales, then the sum of the ten questions indicates the degree of depression. The theoretical score range is from 0 (no depression) to 50 (maximum depression).
  Mild depression: MDI total score from 21 to 25 Moderate depression: MDI total score from 26 to 30 Severe depression: MDI total score of 31 or higher
Fracture risk | Baseline cross sectional data
  FRAX® score. The FRAX® tool has been developed to evaluate fracture risk of patients. It is based on individual patient models that integrate the risks associated with clinical risk factors.
  The FRAX® algorithms give the 10-year probability of fracture. The output is a 10-year probability of hip fracture and the 10-year probability of a major osteoporotic fracture (clinical spine, forearm, hip or shoulder fracture).
Change in Fracture risk | 10 year follow-up
  FRAX® score. The FRAX® tool has been developed to evaluate fracture risk of patients. It is based on individual patient models that integrate the risks associated with clinical risk factors.
  The FRAX® algorithms give the 10-year probability of fracture. The output is a 10-year probability of hip fracture and the 10-year probability of a major osteoporotic fracture (clinical spine, forearm, hip or shoulder fracture).
Obstructive pulmonary disease | Baseline cross sectional data
  Nitric oxide in exhaled breath
Obstructive pulmonary disease | 10 year follow-up
  Change in Nitric oxide in exhaled breath
Prevalence of Peripheral artery disease | Baseline cross sectional data
  Ankle-brachial-index (ABI) is measured using a Doppler meter by determining the systolic pressure in the arm and ankle.
Change in Peripheral artery disease | 10 years follow-up
  Ankle-brachial-index (ABI) is measured using a Doppler meter by determining the systolic pressure in the arm and ankle.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne D Rasmussen, Professor, MD, DMSc, Principal Investigator — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Allan Rasmussen, MD, Study Director — Department of Transplantation and Digestive Diseases, Copenhagen University Hospital - Rigshospitalet; Klaus F Kofoed, Professor, MD, PhD, DMSc, Study Director — Department of Cardiology, Copenhagen University Hospital - Rigshospitalet; Tor Biering-Sørensen, Professor, MD, MSc, PhD, Study Director — Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Suarez-Zdunek MA, Arentoft NS, Krohn PS, Lauridsen EHE, Afzal S, Hogh J, Thomsen MT, Knudsen AD, Nordestgaard BG, Hillingso JG, Villadsen GE, Holland-Fischer P, Rasmussen A, Fialla AD, Feldt-Rasmussen U, Nielsen SD. Prevalence of hyperthyroidism and hypothyroidism in liver transplant recipients and associated risk factors. Sci Rep. 2024 Apr 3;14(1):7828. doi: 10.1038/s41598-024-58544-3. PMID 38570629
- [Derived] Thomsen MT, Hogh J, Knudsen AD, Jensen AMR, Gelpi M, Villadsen GE, Abazi R, Holland-Fischer P, Kober L, Clemmesen O, Krohn PS, Hillingso J, Vilsboll T, Biering-Sorensen T, Kofoed KF, Nordestgaard BG, Rasmussen A, Nielsen SD. The Danish comorbidity in liver transplant recipients study (DACOLT): a non-interventional prospective observational cohort study. BMC Gastroenterol. 2021 Apr 1;21(1):145. doi: 10.1186/s12876-021-01733-5. PMID 33794793